CLINICAL TRIAL: NCT02906358
Title: Evaluating Clinic- and Community-Based Pain Self-Care Programs for Low-Income Hispanics on Opioids
Brief Title: Trial of Chronic Pain Self-Management in Clinic or Community for Low-Income Hispanics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The University of Texas at San Antonio (Other); Bexar County Hospital District DBA University Health System (Other); San Antonio Public Libraries (Unknown); South Central Area Health Education Center (Unknown); The University of Texas System Healthcare Safety & Effectiveness Grants Program (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC20150600H
Record Dates: First submitted 2016-09-07; First posted 2016-09-20 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2017-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Community-based pain self-management (Active Comparator): Community-based pain self-management: two, one-hour meetings monthly for the first three months (6 meetings) and one meeting per month for the last three months (total 9 meetings)
  Interventions: Behavioral: Community-based pain self-management
- Clinic-based pain self-management (Active Comparator): Clinic-based pain self-management: 30-45 minute individualized meetings once monthly for 6 months (total 6 meetings)
  Interventions: Behavioral: Clinic-based pain self-management

INTERVENTIONS:
Behavioral: Community-based pain self-management
  Arms: Community-based pain self-management
Behavioral: Clinic-based pain self-management
  Arms: Clinic-based pain self-management

SUMMARY:
The purpose of this study is to conduct a parallel group, randomized trial of a chronic pain self-management program in clinic or community settings to educate and support low-income, Hispanic patients with chronic pain to adopt evidence-based pain self-care behaviors and activities.

DETAILED DESCRIPTION:
Background and Significance

Over the past two decades, opioid analgesic (OA) drugs have been increasingly prescribed for chronic pain despite little to no effectiveness of treatment >6 months. In prospective cohorts, OA therapy can worsen pain and disability by promoting a sedentary lifestyle. With rapidly rising deaths from OA overdose and the lack of evidence of long-term effectiveness, the U.S. Department of Health and Human Services (HHS) has developed its National Pain Strategy that sharply limits use of OAs and recommends non-pharmacologic interventions as first line approaches to manage chronic pain. A key aspect of a non-pharmacologic approach to managing chronic pain is educating patients about self-management in order to help them lead more productive lives and perform daily activities despite their pain. Self-management training is especially important for low-income patients who need practical, low cost ways to learn how to live fuller, more productive lives despite having chronic pain. To respond to this need to support low-income patients with chronic pain, we developed a chronic pain self-management program based on unmet needs identified by stakeholders from rural, largely Hispanic communities. We conducted a randomized trial to examine outcomes of two settings to deliver this self-management training program. Both settings evaluated whether patients' function improved when the same program was delivered in clinic in individual meetings with a trained community health worker or in a local community-based setting from group lectures by content experts. The training program in both settings offered education and training about such topics as: pain physiology and goal setting; stretching; strengthening; massage, and mindfulness techniques. This program not only reflects the unmet needs of rural, predominantly Hispanic stakeholders with chronic pain but also elements of other self-management programs for patients with chronic back and lower extremity musculoskeletal pain. However, this program was specifically designed for a low literacy, bilingual patient population with limited access to resources to help with non-pharmacologic management of chronic pain.

Objective:

To develop a chronic pain self-management program reflecting community stakeholders' priorities and conduct a randomized trial to evaluate functional outcomes from training in two settings. Subjects will be randomized to receive a 6-month pain self-management training program in: 1) Six 30-to-45 minute individual meetings with a trained community health worker in clinic or 2) nine 1-hour meetings for group lectures by content experts and practicing physical activities held in nearby public libraries.

Study Design:

The investigators conducted a parallel group, randomized trial of clinic- and community-based programs to educate and promote pain self-management among low-income, predominantly Hispanic patients aged 35-70 who had been prescribed at least two months of OA therapy for chronic non-cancer back and lower extremity pain. Patients were recruited from two primary care clinics and one HIV clinic that treat low-income patients. A total of 111 subjects were randomized to: 1) clinic-based meetings one-on-one with a trained community health worker, or 2) a community-based program in a local library with group lectures by content experts and training in exercises. The same low literacy PowerPoint educational program in Spanish or English was presented to both study arms except in the community, eight lectures about chronic pain self-management were presented plus one lecture about using library resources (biweekly for three months then monthly for three months). Whereas, in the clinic arm, the content was condensed to be covered in six monthly 30-45 minute meetings with the community health worker. To increase availability for subjects in the community arm, the same group session was offered twice a week. Sessions included: 1) Orientation to the pain program; 2) Pain physiology exercises/stretching; 3) Stress management and mindfulness; 4) Massage therapy approaches; 5) Nutrition; 6) Sleep hygiene; 7) Relapse prevention; 8) Health literacy (Internet resources); and 9) Review and long-term pain self-management strategies. To keep the group size manageable, the pain self-management program was held in two cohorts to meet library and clinic space limitations.

All subjects received copies of slides from sessions with photos of local Hispanic community members performing stretching and strengthening exercises at different levels of difficulty. Participants also received activity logs to track personal goals, program DVDs (walking exercises, self-massage techniques), exercise mats, tennis balls for massage and multi-pronged self-massage tools. Physical therapy students helped patients select personalized goals for physical activities. All participants received text messages and phone calls from a coordinator (community) or a community health worker (clinic) to review progress and reinforce meeting attendance. Missed sessions were made up with a coordinator (community arm) or a community health worker (clinic arm).

Baseline and follow-up measures were conducted by physical therapy students, CHWs, or team members not involved in that study arm. Twelve measures of physical, cognitive, and psychological, function and pain were assessed at 6 months in the clinic or the community location and 6 of these were also assessed at 3 months. The primary outcome measure was the five times sit-to-stand test (5XSTS) that was assessed at both 3 and 6 months and reflects both lower extremity strength and balance. The 5XSTS is significantly associated with disability and risk of falls. Secondary outcomes include: 6-minute distance walk test (6MW); Borg Perceived Effort test (Borg effort); 50-foot speed walk test (50FtSW); 12-Item Short Form Survey Physical Component Summary (SF-12 PCS); and Patient Specific Functional Scale (PSFS). Measures of psychological function include: 12-Item Short Form Survey Mental Component Summary (SF-12 MCS), Brief Pain Inventory (BPI), Patient Health Questionnaire-9 (PHQ-9) and the Tampa Scale for Kinesiophobia (TSK). To assess cognitive function, the Symbol-Digit Modalities Test (SDMT) evaluates attention and psychomotor speed. All measures were performed at baseline and the 6-month study endpoint except the following measures also assessed at three months: 5XSTS, 50FtSW, BPI, PSFS and SDMT. These are all validated functional measures (see below). The practical self-management training program evaluated in this trial may offer a valuable resource for primary care practices striving to support their patients with chronic pain, especially those with limited access to other resources.

Impact:

If either or both of the approaches to deliver this chronic pain self-management training program improve patient functional outcomes, they can be easily replicated to evaluate in other low-income populations to improve function and possibly even reduce dependence on OA therapy.

ELIGIBILITY:
Inclusion Criteria:

* Active patient in two study primary care clinics or HIV clinic in same system
* Prescribed OAs >2 mos in the past year
* Back/lower extremity pain
* English or Spanish speaking

Exclusion Criteria:

* Unstable comorbidity
* Cardiovascular/pulmonary disease that prevents exercise
* Cancer-related pain
* Significant mental health disorder
* Alcohol or drug abuse
* Inability to walk unassisted for at least one block
* Inability to provide consent (e.g., dementia)
* Residing more than 10 miles from clinic (poor transportation)
* Patients who are unable or unwilling to attend clinic- or community-based sessions

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Turner, MD, Principal Investigator — UT Health Science Center at San Antonio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou R, Turner JA, Devine EB, Hansen RN, Sullivan SD, Blazina I, Dana T, Bougatsos C, Deyo RA. The effectiveness and risks of long-term opioid therapy for chronic pain: a systematic review for a National Institutes of Health Pathways to Prevention Workshop. Ann Intern Med. 2015 Feb 17;162(4):276-86. doi: 10.7326/M14-2559. PMID 25581257
- [Background] Jensen MK, Thomsen AB, Hojsted J. 10-year follow-up of chronic non-malignant pain patients: opioid use, health related quality of life and health care utilization. Eur J Pain. 2006 Jul;10(5):423-33. doi: 10.1016/j.ejpain.2005.06.001. Epub 2005 Jul 28. PMID 16054407
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893
- [Background] French DJ, France CR, Vigneau F, French JA, Evans RT. Fear of movement/(re)injury in chronic pain: a psychometric assessment of the original English version of the Tampa scale for kinesiophobia (TSK). Pain. 2007 Jan;127(1-2):42-51. doi: 10.1016/j.pain.2006.07.016. Epub 2006 Sep 7. PMID 16962238
- [Background] Woby SR, Roach NK, Urmston M, Watson PJ. Psychometric properties of the TSK-11: a shortened version of the Tampa Scale for Kinesiophobia. Pain. 2005 Sep;117(1-2):137-44. doi: 10.1016/j.pain.2005.05.029. PMID 16055269
- [Background] Simmonds MJ, Ortega C, Simmonds KP. Pain, Emotion and Cognition. ln: Pickering G, Gibson S, eds. Switzerland: Springer International Publishing; c2015. Chapter 11, Physical Therapy and Exercise: Impacts on Pain, Mood, Cognition, and Function; p. 167-186.
- [Background] Smith A. Symbol Digits Modalities Test. Western Psychological Services: Los Angeles, 1982.
- [Background] Valerio MA, Rodriguez N, Winkler P, Lopez J, Dennison M, Liang Y, Turner BJ. Comparing two sampling methods to engage hard-to-reach communities in research priority setting. BMC Med Res Methodol. 2016 Oct 28;16(1):146. doi: 10.1186/s12874-016-0242-z. PMID 27793191
- [Background] Butler DS, Moseley GL. Explain Pain. Adeliade, South Australia: Noigroup Publications; 2013.
- [Background] Jones SE, Kon SS, Canavan JL, Patel MS, Clark AL, Nolan CM, Polkey MI, Man WD. The five-repetition sit-to-stand test as a functional outcome measure in COPD. Thorax. 2013 Nov;68(11):1015-20. doi: 10.1136/thoraxjnl-2013-203576. Epub 2013 Jun 19. PMID 23783372
- [Background] Steffen TM, Hacker TA, Mollinger L. Age- and gender-related test performance in community-dwelling elderly people: Six-Minute Walk Test, Berg Balance Scale, Timed Up & Go Test, and gait speeds. Phys Ther. 2002 Feb;82(2):128-37. doi: 10.1093/ptj/82.2.128. PMID 11856064
- [Background] Smeets RJ, Hijdra HJ, Kester AD, Hitters MW, Knottnerus JA. The usability of six physical performance tasks in a rehabilitation population with chronic low back pain. Clin Rehabil. 2006 Nov;20(11):989-97. doi: 10.1177/0269215506070698. PMID 17065542
- [Background] Bohannon RW. Test-retest reliability of the five-repetition sit-to-stand test: a systematic review of the literature involving adults. J Strength Cond Res. 2011 Nov;25(11):3205-7. doi: 10.1519/JSC.0b013e318234e59f. PMID 21904240
- [Background] Ware JE, Kosinski M, Keller SD. SF-12: How to Score the SF-12 Physical and Mental Health Summary Scales. 2nd ed. Boston: The Health Institute; 1995.
- [Background] Abbott JH, Schmitt J. Minimum important differences for the patient-specific functional scale, 4 region-specific outcome measures, and the numeric pain rating scale. J Orthop Sports Phys Ther. 2014 Aug;44(8):560-4. doi: 10.2519/jospt.2014.5248. Epub 2014 May 14. PMID 24828475
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Derived] Turner BJ, Rodriguez N, Bobadilla R, Hernandez AE, Yin Z. Chronic Pain Self-Management Program for Low-Income Patients: Themes from a Qualitative Inquiry. Pain Med. 2020 Feb 1;21(2):e1-e8. doi: 10.1093/pm/pny192. PMID 30312459
- [Derived] Turner BJ, Liang Y, Simmonds MJ, Rodriguez N, Bobadilla R, Yin Z. Randomized Trial of Chronic Pain Self-Management Program in the Community or Clinic for Low-Income Primary Care Patients. J Gen Intern Med. 2018 May;33(5):668-677. doi: 10.1007/s11606-017-4244-2. Epub 2018 Jan 3. PMID 29299814
- See also: Department of Health and Human Services: ASPE Issue Brief. Opioid Abuse in the U.S. and HHS Actions to Address Opioid-Drug Related Overdoses and Deaths — http://aspe.hhs.gov/sp/reports/2015/OpioidInitiative/ib_OpioidInitiative.pdf
- See also: The Progressive Goal Attainment Program (PGAP®). An Evidence-Based Treatment Program for Reducing Disability Associated with Pain, Depression, Cancer and other Chronic Health Conditions. — http://www.pgapworks.com/en/whatisthepgap/index.php
- See also: Moore P, Cole F. The Pain Toolkit. — http://www.paintoolkit.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Community-based Pain Self-management: Community-based pain self-management: two, one-hour meetings monthly for the first three months (6 meetings) and one meeting per month for the last three months (total 9 meetings)
  Community-based pain self-management
- Clinic-based Pain Self-management: Clinic-based pain self-management: 30-45 minute individualized meetings once monthly for 6 months (total 6 meetings)
  Clinic-based pain self-management
Period: Overall Study
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Started | 58 | 53
Completed 3 Month Measures | 36 | 33
Completed (Includes participants who completed the entire program and 6 month measures) | 36 | 31
Not Completed | 22 | 22
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Lost to Follow-up | 12 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management | Total
Number analyzed (Participants) | 58 | 53 | 111
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (8.7) | 56.2 (9.4) | 56.5 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 24 | 61
  Male | 21 | 29 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 45 | 42 | 87
  Non-Hispanic White | 8 | 6 | 14
  Non-Hispanic Black | 5 | 5 | 10
Primary Language [Count of Participants; unit: Participants]
  English | 45 | 36 | 81
  Spanish | 13 | 17 | 30
Marital Status [Count of Participants; unit: Participants]
  Married | 18 | 16 | 34
  Other (single, divorced, separated, widowed) | 40 | 37 | 77
Employment Status [Count of Participants; unit: Participants]
  Employed | 6 | 1 | 7
  Unemployed (retired, disabled, unemployed) | 52 | 52 | 104
Insurance Type [Count of Participants; unit: Participants]
  Private Insurance | 4 | 6 | 10
  Medicare | 21 | 17 | 38
  Medicaid | 13 | 11 | 24
  Unisured | 20 | 19 | 39
BMI [Mean (Standard Deviation); unit: kg/m^2] | 35.5 (8.0) | 33.3 (8.8) | 34.5 (8.4)
Pain Location [Count of Participants; unit: Participants]
  Neck | 0 | 3 | 3
  Upper Extremity | 3 | 1 | 4
  Back | 19 | 13 | 32
  Abdomen | 1 | 0 | 1
  Lower Extremity | 5 | 4 | 9
  Multiple areas | 30 | 32 | 62

OUTCOME MEASURES:

1. Primary Outcome: Five Times Sit-to-stand (5XSTS)
Description: Participants are instructed to sit and stand up five times as fast as they can from a standard armless chair while the researcher times how many seconds it takes them to complete the task. After a brief rest, they repeat the test a second time and the average of two tests is calculated.
Time Frame: Change from Baseline sit-to-stand at 3 and 6 months
Population: We report a completers analysis of unadjusted change in outcome measures in community and clinic arms at 3 months (for selected measures) and 6 months (for all measures), that include only completers in the participant flowchart (Community arm=36, Clinic arm 3 months=33, 6 months=31). Completers may differ by outcome if data was missing.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
seconds
  Change from Baseline Score at 3 Months: number analyzed (Participants) | 35 | 32
  Change from Baseline Score at 3 Months | -4.53 (6.78) | -5.20 (17.53)
  Change from Baseline Score at 6 Months: number analyzed (Participants) | 32 | 30
  Change from Baseline Score at 6 Months | -4.18 (6.45) | -6.43 (14.11)

2. Secondary Outcome: 50-foot Speed Walk (50FtSW)
Description: This test requires participants to walk along a 25-foot walkway turn around and return to the starting point. They are instructed to safely walk as fast as they can and the time taken to complete the test is recorded in seconds.
Time Frame: Change from Baseline 50-foot speed walk at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
seconds
  Change from Baseline Score at 3 Months | -1.58 (5.55) | -1.22 (4.29)
  Change from Baseline Score at 6 Month: number analyzed (Participants) | 36 | 31
  Change from Baseline Score at 6 Month | -1.32 (7.16) | -1.42 (4.85)

3. Secondary Outcome: Patient Specific Functional Scale (PSFS)
Description: This is a brief, one-page document that prompts subjects to identify limitations to three activities, rank the importance of these activities, and track progress over time. The activities are scored on a scale of 0 to 10, where 0 indicates that the subject is unable to perform the activity and 10 indicates ability to perform the activity at the same level as before the injury or problem. The total summed score is divided by the number of activities, where a lower score would indicate less ability to perform the task, and the higher score would indicate easier performance of the task.
Time Frame: Change from Baseline PSFS at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
units on a scale
  Change from Baseline Score at 3 Months: number analyzed (Participants) | 36 | 32
  Change from Baseline Score at 3 Months | 1.07 (1.95) | 1.04 (1.66)
  Change from Baseline Score at 6 Months: number analyzed (Participants) | 36 | 30
  Change from Baseline Score at 6 Months | 1.64 (2.28) | 1.65 (1.77)

4. Secondary Outcome: Symbol-Digit Modalities Test (SDMT)
Description: Participants refer to a key on top of a page to translate non-verbal symbols to an alpha-numeric digit. The participants then fill in boxes (written and oral versions) with the correct digit assigned to a particular symbol. Total correct responses within 90 seconds were measured. The score of the test is the number of correct substitutions completed within the time limit, with a maximum score of 110. A score under 33 is generally considered to be a clear indicator of the existence of some type of cognitive disorder. The higher the score, the better the cognitive function.
Time Frame: Change from Baseline SDMT at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
units on a scale
  Change from Baseline Score at 3 Months: number analyzed (Participants) | 36 | 32
  Change from Baseline Score at 3 Months | 4.19 (6.61) | 6.84 (10.0)
  Change from Baseline Score at 6 Month: number analyzed (Participants) | 36 | 30
  Change from Baseline Score at 6 Month | 4.61 (8.67) | 7.37 (8.94)

5. Secondary Outcome: The Brief Pain Inventory (BPI): Severity
Description: The BPI is brief and uses simple 0-10 rating scales to measure pain intensity, where zero is no pain and ten is most intense pain imaginable.
Time Frame: Change from Baseline BPI at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
units on a scale
  Change from Baseline Score at 3 Months | -0.90 (1.59) | -1.17 (2.00)
  Change from Baseline Score at 6 Month: number analyzed (Participants) | 36 | 31
  Change from Baseline Score at 6 Month | -0.95 (1.84) | -1.08 (2.09)

6. Secondary Outcome: The Brief Pain Inventory (BPI): Interference
Description: The BPI is brief and uses simple 0-10 rating scales to measure the degree to which pain interferes with common dimensions of feeling and function, where zero is does not interfere and ten is completely interferes.
Time Frame: Change from Baseline BPI at 3 and 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 33
units on a scale
  Change from Baseline Score at 3 Months | -0.31 (1.84) | -1.15 (4.10)
  Change from Baseline Score at 6 Months: number analyzed (Participants) | 36 | 31
  Change from Baseline Score at 6 Months | -1.09 (2.46) | -1.37 (2.42)

7. Secondary Outcome: 6-minute Distance Walk (6MW)
Description: For this test, participants walk as far as they can for six minutes, and the total distance in feet is measured with a surveyor's wheel pushed by a research assistant walking behind the subject. Participants can pause or stop as necessary.
Time Frame: Change from Baseline 6-minute distance walk at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 34 | 31
feet | 20.0 (291.9) | 193.9 (429.0)

8. Secondary Outcome: Borg Perceived Effort (Borg)
Description: Completed in conjunction with the 6-minute walk, this measures intensity and perceived effort after the test using a 0-10 Likert-type scale. Anchor words for the effort scales are "no effort" and "most intense effort imaginable."
Time Frame: Change from Baseline perceived effort at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 34 | 29
units on a scale | -0.21 (3.60) | -1.76 (4.19)

9. Secondary Outcome: Medical Outcomes Study 12-Item Short Form Physical Component Summary (SF-12 PCS)
Description: The 12-item Short Form Health Survey created for Medical Outcomes Study measures physical summary scores through a brief survey with limited respondent burden while retaining precision. Physical Health Composite Scores are computed using the scores of 12 questions and range from 0 to 100, where 0 indicates the lowest level of health, and 100 indicates the highest level of health.
Time Frame: Change from Baseline SF-12 PCS at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 35 | 30
units on a scale | 2.20 (8.56) | 6.76 (9.99)

10. Secondary Outcome: Medical Outcomes Study 12-Item Short Form Mental Component Summary (SF-12 MCS)
Description: The 12-item Short Form Health Survey created for Medical Outcomes Study measures mental summary scores through a brief survey with limited respondent burden while retaining precision. Mental Health Composite Scores are computed using the scores of 12 questions and range from 0 to 100, where 0 indicates the lowest level of mental health, and 100 indicates the highest level of mental health.
Time Frame: Change from baseline SF-12 MCS at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 35 | 30
units on a scale | 41.44 (12.58) | 39.39 (12.3)

11. Secondary Outcome: Patient Health Questionnaire -9 (PHQ-9)
Description: The PHQ-9 is a brief, self-administered questionnaire that assesses somatic symptom severity. Participants rate the severity of 15 somatic symptoms as 0 (not bothered at all), 1 (bothered a little) or 2 (bothered a lot). The scores are totaled, with a possible total of 30, which would mean the most severe somatic symptoms, and 0 meaning the least somatic symptoms.
Time Frame: Change from Baseline PHQ-9 at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 31
units on a scale | -2.08 (6.42) | -3.45 (6.81)

12. Secondary Outcome: Tampa Scale for Kinesiophobia (TSK)
Description: This is a 11-item questionnaire, where individuals score items on a scale of 1 to 4 (1=strongly disagree, 4=strongly agree) to measures fear of completing physical activities. The scores are totaled for all items, to give a possible score of 44, which would indicate a greater fear of injuring oneself. A lower score would indicate less fear of injury to oneself.
Time Frame: Change from Baseline TSK at 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
Number analyzed (Participants) | 36 | 31
units on a scale | -2.64 (6.32) | -2.77 (7.10)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for 11 months, the duration of the program.
Groups:
- Community-based Pain Self-management: Community-based pain self-management: two, one-hour monthly meetings for first three months (6 meetings) and one meeting per month for the last three months (total 9 meetings)
  Community-based pain self-management
Arm/Group | Community-based Pain Self-management | Clinic-based Pain Self-management
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/53
Serious Adverse Events (participants affected / at risk) | 3/58 | 0/53
Other Adverse Events (participants affected / at risk) | 3/58 | 2/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community-based Pain Self-management (N=58) | Clinic-based Pain Self-management (N=53)
Fractured leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fractured their leg after missing a step while entering the house during a family gathering.
Gout attack (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient went to the hospital for heart attack symptoms and was told he had gout.
Diabetic foot infection leading to leg amputation (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient had neuropathy and uncontrolled diabetes which caused a leg amputation.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community-based Pain Self-management (N=58) | Clinic-based Pain Self-management (N=53)
Sprained wrist (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient wore a wrist brace and stated that they have had wrist problems and occasionally use the brace when they have discomfort.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell while walking inside home after sitting outside with family, a daily routine.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell back after getting up from a chair in the kitchen.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Patient fell at the grocery store which she stated has happened previously because of problems with balance.
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Patient fell at home before the program had started.

LIMITATIONS AND CAVEATS:
Limitations of our study include the absence of a control group to gain clinic support, unanticipated adverse events, challenges recruiting and retaining subjects, lack of long-term follow-up and possible lack of generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes